CLINICAL TRIAL: NCT04005794
Title: Physiology-based Virtual Reality Training for Social Skills in Schizophrenia
Brief Title: Virtual Reality Training for Social Skills in Schizophrenia - Comparison With Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Sohee Park, Professor of Psychology, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MH106748-R33
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Social Skills
Keywords: schizophrenia; social skills training; social brain network; virtual reality; simulation; functional outcome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Social Skills | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Two conditions are compared in individuals with schizophrenia in a cross over design: social skills Virtual Reality (VR) training and active control condition of cognitive training game (non-social, cognitive video game).
  Participants are assigned at random to either start with social VR (Virtual Reality) skills training and cross over to the cognitive game at baseline, or start with the cognitive game and cross over to the social VR (Virtual Reality) training. They are assessed at baseline for symptoms, social function, emotion perception.
  They participate in the assigned condition until completion. They then get post-training assessments after which they switch over to the other condition.
  This cross-over design was implemented due to the closure of the laboratory during the pandemic.
  Healthy controls are run on the baseline tasks to provide the comparison data for the patient groups but the controls do not undergo VR training nor they yield any clinical symptoms data.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to the training condition. Schizophrenia participants know which games they are playing so although we do not tell them whether they are being trained for social skills or not, it is not possible to make sure that they are unaware of the types of games that they are asked to play
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizophrenia group (Experimental): Participants undergo both social VR (virtual reality) training and a control game sequentially. They are randomly assigned at baseline to one training condition. After completing 8 sessions, they cross over to the other condition. There are two training conditions: social VR and cognitive training game.
  Interventions: Behavioral: social VR (virtual reality) training; Behavioral: Cognitive training (control game)
- Healthy Controls (No Intervention): Healthy controls are recruited to yield comparison data. They do not undergo training.

INTERVENTIONS:
Behavioral: social VR (virtual reality) training — Social skills game that we developed in the R21 phase will be used across 8 sessions of training in the lab. Each session is about 1 hour long. Participants come to the lab twice a week for 4-5 weeks.
  Arms: Schizophrenia group
Behavioral: Cognitive training (control game) — Commercially available cognitive training program will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games.
  Arms: Schizophrenia group

SUMMARY:
Social impairments are core features of schizophrenia that lead to poor outcome. Social skills and competence improve quality of life and protect against stress-related exacerbation of symptoms, while supporting resilience, interpersonal interactions, and social affiliation. To improve outcome, it is necessary to remediate social deficits. Existing psychosocial interventions are moderately effective but the effort-intensive nature (high burden), low adherence, and weak transfer of skills to everyday life present significant hurdles toward recovery. Thus, there is a dire need to develop effective, engaging and low-burden social interventions for people with schizophrenia that will result in better compliance rates and functional outcome.

In a previous pilot study, the investigators tested the effectiveness of a novel adaptive virtual reality (VR) intervention in improving targeted social cognitive function (social attention, as indexed by eye scanning patterns) in individuals with schizophrenia. 10 sessions of 1-hour VR intervention were sufficient to engage the target mechanism of social attention and improve negative symptoms. Acceptability and compliance were very high among the participants. In fact, improvements were seen at about 4-5 sessions. Therefore, we used 8 sessions for the R33 phase.

The next phase, supported by a R33 grant compares the VR social skills training with a control condition. This new protocol includes a control condition for the exposure to computerized training across the 8 sessions and incidental exposure to social interactions (i.e. interactions with experimenters twice a week for 4-5 weeks). The control condition consists of commercially available cognitive video games played on the same computer for the same duration as the social VR training condition. This control condition is called Cognitive training game condition.

DETAILED DESCRIPTION:
The effectiveness of the social skills VR training at an optimal dose will be compared with an active control condition (computerized cognitive training game) in improving social attention (Social Engagement Latency: SEL), symptoms and social cogitive functioning in a pilot randomized cross-over trial.

Participants with schizophrenia will undergo a baseline assessment of social cognitive functioning, and clinical symptoms. Potential changes after Social skills VR training compared with cognitive game training will be examined.

Individuals with schizophrenia will be randomized to either the social skills VR training or the cognitive training at baseline. They will then participate in 8 sessions of social skills VR training or cognitive training (1 hour per session, twice a week for 4-5 weeks). After completion of the 8 sessions per training condition, they will cross over and participate in the other condition.

Social engagement latency (SEL) will be used as a measure of social attention which is the primary target. The Social Functional Scale (Birchwood, 1991), the the Scale for the Assessment of Negative Symptoms (SANS) and the Scale for the Assessment of Positive Symptoms (SAPS) will be used to assess social functioning and symptoms. Emotion perception will be assesed by the Bell-Lysaker Emotion Recognition Task (BLERT-A).

Matched healthy control participants will be recruited to obtain comparison data for optimal performance levels but these healthy control participants will not undergo social skills training.

Lastly, at the end of the R33 project, if this VR social skills VR training shows that it can improve social attention, which may improve social outcome in schizophrenia, it will be possible to refine the protocol to make the method more accessible, less burdensome and widely available in the future by moving towards a mobile application.

ELIGIBILITY:
1. Inclusion and Exclusion Criteria for Individuals with Schizophrenia:

   Inclusion criteria for schizophrenia group:
   * Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) Axis 1 Diagnosis of schizophrenia
   * Wechsler Abbreviated Scale of Intelligence (WASI) intelligence quotient (IQ) > 85
   * Currently taking antipsychotic medication
   * No change in current psychotropic medications or housing within the past 30 days. Those patients whose medication or housing situation has changed within a month, we will wait list them until their situation stabilizes.

   Exclusion criteria for schizophrenia group:
   * Diagnostic and Statistical Manual of Mental Disorders-5 (DSM 5) Axis 1 diagnosis other than schizophrenia
   * Diagnosed organic brain disease, brain lesions, history of head traumas, neurological disorders or other conditions that involve the degeneration of the central nervous system (e.g. multiple sclerosis)
   * Substance/alcohol dependence during the past 1 year
   * Tardive dyskinesia
2. Inclusion and Exclusion Criteria for Healthy Control Participants:

   * Wechsler Abbreviated Scale of Intelligence (WAIS) IQ > 85
   * No Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) Axis 1 diagnosis of psychotic disorders in themselves or their families (e.g. schizophrenia, bipolar disorder).
   * No antipsychotic medications
   * No diagnosed organic brain disease, brain lesions, history of head traumas, neurological disorders or other conditions that involve the degeneration of the central nervous system (e.g. multiple sclerosis)
   * No substance/alcohol dependence during the past 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sohee Park, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
We are comparing a social skills game in virtual reality with a cognitive training software. After the study is completed, we will make the protocol and the methods available to all those who request this information.
Supporting Information: Study Protocol
Time Frame: After the study has ended and we have been able to publish the outcome of the study. This is expected to be within 2 years of the completion of the study.
Access Criteria: Interested parties should contact the P.I. by email.

REFERENCES:
- [Result] Adery LH, Ichinose M, Torregrossa LJ, Wade J, Nichols H, Bekele E, Bian D, Gizdic A, Granholm E, Sarkar N, Park S. The acceptability and feasibility of a novel virtual reality based social skills training game for schizophrenia: Preliminary findings. Psychiatry Res. 2018 Dec;270:496-502. doi: 10.1016/j.psychres.2018.10.014. Epub 2018 Oct 9. PMID 30326433
- [Result] Torregrossa LJ, Bian D, Wade J, Adery LH, Ichinose M, Nichols H, Bekele E, Sarkar N, Park S. Decoupling of spontaneous facial mimicry from emotion recognition in schizophrenia. Psychiatry Res. 2019 May;275:169-176. doi: 10.1016/j.psychres.2019.03.035. Epub 2019 Mar 20. PMID 30921747
- [Result] Wade J, Nichols HS, Ichinose M, Bian D, Bekele E, Snodgress M, Amat AZ, Granholm E, Park S, Sarkar N. Extraction of Emotional Information via Visual Scanning Patterns: A Feasibility Study of Participants with Schizophrenia and Neurotypical Individuals. ACM Trans Access Comput. 2018 Nov;11(4):23. doi: 10.1145/3282434. PMID 30627303

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Schizophrenia patients undergo both Social VR training and Cognitive Training
Groups:
- Social Skills VR (Virtual Reality) Training, Then Cognitive Training: 1. social skills VR training: Social skills game that we developed in the R21 phase will be used across 8 sessions of training in the lab. Each session is about 1 hour long. Participants come to the lab twice a week for 4-5 weeks.
  2. Cognitive Training: Commercially available cognitive training program will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games. They complete 8 sessions over 4-5 weeks
- Cognitive Training, Then VR Social Skills Training: 1. Cognitive Training: Commercially available cognitive training program will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games. They complete 8 sessions over 4-5 weeks.
  2. VR social skills training: Social skills game that we developed in the R21 phase will be used across 8 sessions of training in the lab. Each session is about 1 hour long. Participants come to the lab twice a week for 4-5 weeks.
Period: Overall Study
Arm/Group | Social Skills VR (Virtual Reality) Training, Then Cognitive Training | Cognitive Training, Then VR Social Skills Training | Healthy Controls
Started (We started recruiting and enrolling participants in Oct 15, 2021) | 11 | 11 (Started Oct 15, 2021.) | 28 (Started Oct 15 2021)
Completed | 11 | 7 (Study completes in May 2024) | 28 (Study completed in May 2024)
Not Completed | 0 | 4 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: There were 22 in the schizophrenia group. 11 began with the social VR training followed by cognitive training game. The other 11 began with cognitive game and then cross over-ed to the social vr training.
  Healthy participants do not train.
Groups:
- Social Skills VR Training, Then Cognitive Training Game: 1. Social skills VR training: Social skills VR game that we developed in the R21 phase will be used across 8 sessions of training in the lab. Each session is about 1 hour long. Participants come to the lab twice a week for 4-5 weeks.
  2. Cognitive Training Game: Commercially available cognitive training program will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games. They complete 8 sessions over 4-5 weeks.
- Cognitive Training Game, Then Social Skills VR Training: 1. Cognitive Training Game: Commercially available cognitive training program will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games. They complete 8 sessions over 4-5 weeks
  2. Social skills VR training: Social skills VR game that we developed in the R21 phase will be used across 8 sessions of training in the lab. Each session is about 1 hour long. Participants come to the lab twice a week for 4-5 weeks.
- Healthy Controls: Healthy controls are recruited to yield comparison data. They do not undergo training.
  They are not interviewed for clinical symptoms
- Total: Total of all reporting groups
Arm/Group | Social Skills VR Training, Then Cognitive Training Game | Cognitive Training Game, Then Social Skills VR Training | Healthy Controls | Total
Number analyzed (Participants) | 11 | 11 | 28 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.74 (12.58) | 45.39 (11.16) | 33.43 (15.35) | 40.50 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 15 | 19
  Male | 9 | 9 | 13 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 10 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 9 | 4 | 20
  White | 3 | 2 | 11 | 16
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 28 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Social Attention: Social Engagement Latency (SEL)
Description: Social engagement latency is defined as the time taken to select an avatar in the social skills training game.
  Social engagement latency is measured in milliseconds. We report the difference in SEL at post training from baseline for Sz group only
Time Frame: Baseline and social VR post-training (after 8 sessions)
Population: We examined the social engagement for the social VR game condition only. Commercially available cognitive games did not have a social component and therefore, they do not yield SEL data. Healthy CO do not participate in any training so they do not yield SEL data
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- VR Social Skills Training: VR social skills training: Social skills game that we developed in the R21 phase will be used across 8 sessions of training in the lab. Each session is about 1 hour long. Participants come to the lab twice a week for 4-5 weeks.
- Cognitive Training: Cognitive Training: Commercially available cognitive training program will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games. They complete 8 sessions over 4-5 weeks
- Healthy Control: Healthy controls are recruited to yield comparison data. They do not undergo training.
Arm/Group | VR Social Skills Training | Cognitive Training | Healthy Control
Number analyzed (Participants) | 18 | 0 | 0
milliseconds | -195 (5.60) |  |
Statistical Analysis 1: Comparison: VR Social Skills Training; Test type: Other; p = 0.004, t-test, 2 sided — Social latency t = 3.215

2. Secondary Outcome: Change in Social Emotion Recognition: Bell-Lysaker Emotion Recognition Task Adult (BLERT-A)
Description: Change in social cognition using the Bell-Lysaker Emotion Recognition Task Adult (BLERT-A). There are 21 videos shown to participants and are scored as either correct (1) or incorrect (0). A total score is provided and can range from 0 to 21, with higher scores indicating a higher social cognition ability, a better outcome.
Time Frame: Baseline and after 8 sessions of social VR training and after 8 sessions of cognitive training game
Population: Patients with schizophrenia participated in both social skills VR game and the cognitive training game. 22 people started but only 18 completed both training. Healthy control participants were tested once at baseline
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Social VR Training: Participants undergo both social VR training and a control game sequentially. They are randomly assigned at baseline to one training condition. After completing 8 sessions, they cross over to the other condition. There are two training conditions: social VR and control game.
  VR social skills training: Social skills game that we developed in the R21 phase will be used across 8 sessions of training in the lab. Each session is about 1 hour long. Participants come to the lab twice a week for 4-5 weeks.
  Cognitive training (control game): Commercially available cognitive training program will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games.
- Cognitive Training Game: Participants play commercially available cognitive training game for 8 sessions. This is a control condition for the social skills VR game.
Arm/Group | Social VR Training | Cognitive Training Game | Healthy Controls
Number analyzed (Participants) | 18 | 18 | 28
score on a scale
  Baseline | 12.68 (0.98) | 12.68 (0.98) | 18 (0.43)
  After Training: number analyzed (Participants) | 18 | 18 | 0
  After Training | 13.00 (1.15) | 13.16 (4.88) |
Statistical Analysis 1: Comparison: Social VR Training vs Cognitive Training Game vs Healthy Controls; Test type: Other; p = 0.213, ANOVA

3. Secondary Outcome: Change in Scale for the Assessment of Negative Symptoms (SANS)
Description: SANS is a 25-item clinical symptom rating scale. It consists subscales of alogia, affective blunting, avolition-apathy, anhedonia-asociality, and attentional impairment. (Andreasen, 1983). Each item is scored on likert scale of 0 (none) to 5 (severe - worse outcome). Total score is summed (range 0-125) with higher scores being a worse outcome Andreasen NC: Scale for the Assessment of Negative Symptoms (SANS) . Iowa City, University of Iowa, 1983
Time Frame: Baseline and after 8 sessions of training for social VR and after 8 sessions of active control game for the schizophrenia group only. CO do not undergo clinical symptoms interview.
Population: This is a clinical interview to assess psychotic symptoms. Therefore healthy control group is not interviewed.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Social VR Training: Severity of symptoms are compared between VR social skills training against the baseline scores
- Cognitive Training Game: Severity of symptoms are compared between cognitive training against the baseline scores
- Healthy Controls: Control participant are not interviewed for psychotic symptoms so there is no data
Arm/Group | Social VR Training | Cognitive Training Game | Healthy Controls
Number analyzed (Participants) | 18 | 18 | 0
score on a scale
  Baseline SANS score | 44.63636364 (3.145494582) | 44.63636364 (3.145494582) |
  After training SANS score | 34.79 (3.287917761) | 43.67 (3.10175999) |
Statistical Analysis 1: Comparison: Social VR Training vs Cognitive Training Game; Test type: Other; p = 0.01, ANOVA

4. Secondary Outcome: Change in Scale for the Assessment of Positive Symptoms (SAPS)
Description: SAPS has 34-items that evaluate hallucinations, delusions, formal thought disorder and bizarre behavior (Andreasen, 1984). Each subscale has a single global score item to rate the overall severity of each symptom domain. Each item is rated for severity from least (0) to most severe (5). Total scores are summed and range from 0-170 with higher scores indicating a worse outcome.
  Andreasen NC: Scale for the Assessment of Positive Symptoms (SAPS) . Iowa City, University of Iowa, 1984. (NC Andreasen - The British Journal of Psychiatry, 1989)
Time Frame: Baseline and after 8 sessions of training for social VR and after 8 sessions of active control game
Population: Healthy controls are not interviewed for clinical symptoms because they are not diagnosed.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Social VR Training: Severity of symptoms are compared between VR social skills training and control game condition against the baseline scores
- Healthy Controls: CO group is not interviewed on clinical symptoms because they do not have the diagnosis of schizophrenia
Arm/Group | Social VR Training | Cognitive Training Game | Healthy Controls
Number analyzed (Participants) | 18 | 18 | 0
score on a scale
  Baseline | 37.86363636 (4.145) | 37.86363636 (4.145) |
  After Training | 28.32 (4.776) | 31.28 (4.008) |
Statistical Analysis 1: Comparison: Social VR Training vs Cognitive Training Game; Test type: Other; p = 0.004, ANOVA

5. Secondary Outcome: Change in Social Outcome: Social Functioning Scale.
Description: Social Functioning Scale (SFS; Birchwood, 1990). SFS consists of 79 items (7 subscales). We use the full scale score. Minimum score is 0 (worst social functioning) and maximum score is 135 (best)
Time Frame: Baseline and after 8 sessions of training for social VR and after 8 sessions of active control game
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Healthy Controls: Healthy controls are recruited to yield comparison data. They do not undergo training.
  Therefore, only baseline scores are available
Arm/Group | Social VR Training | Cognitive Training Game | Healthy Controls
Number analyzed (Participants) | 18 | 18 | 28
score on a scale
  Baseline | 96.63636364 (1.848) | 96.63636364 (1.848) | 107.25 (1.89)
  After training: number analyzed (Participants) | 18 | 18 | 0
  After training | 98.74 (1.849) | 97.56 (1.856) |
Statistical Analysis 1: Comparison: Social VR Training vs Cognitive Training Game vs Healthy Controls; Test type: Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Baseline up to seven months.
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time the consent was signed through participant completion
Groups:
- Social VR Skills Training: 1. Social VR skills training: Social skills game will be used across 8 sessions of training in the lab. Each session is about 1 hour long. They come to the lab twice a week.
- Cognitive Training: 2. Cognitive training: Commercially available cognitive training games will be used to control for the time spent in the lab and associated social interactions as well as the total exposure to computerized games. 8 session across 4-5 weeks
Arm/Group | Social VR Skills Training | Cognitive Training | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/28
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT04005794/Prot_SAP_000.pdf